CLINICAL TRIAL: NCT06700733
Title: Polyetheretherketone (PEEK) Versus Titanium Frameworks for All-on-4 Implant Full-arch Prosthesis: Within-patient Evaluation of Patient Satisfaction, Oral Health-related Quality of Life (OHRQoL), Chewing Efficiency and Maximum Bite Force
Brief Title: PEEK Vs Titanium for All-on-4 Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Khloud Ezzat, lecturer, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0508024RP
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Satisfaction, Patient; Bite Force
Keywords: PEEK; Titanium; All-on-4
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: All selected patients will receive maxillary complete dentures and mandibular screw-retained prosthesis either from PEEK or Titanium framework in a crossover design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): The first 9 patients will receive the PEEK prosthesis (PP) first. After 3 months, chewing efficiency, maximum bite force, patient satisfaction, and OHRQoL will be measured, and PP will be replaced by a Titanium prosthesis (TP). After another 3 months, the measurements will be repeated.
  Interventions: Device: PEEK prosthesis; Device: Titanium prosthesis
- study group 1 (Experimental): The second 9 patients will receive TP first, and after 3 months, measurements will be made. Then, TP was replaced by PP, and measurements will be repeated after another 3 months. This randomization will be made to reduce the effect of prosthesis type and bias
  Interventions: Device: PEEK prosthesis; Device: Titanium prosthesis

INTERVENTIONS:
Device: PEEK prosthesis — For the PP, The PEEK framework will be constructed, the fit of the PEEK framework will be verified intraorally, and the final screw-retained prosthesis will be constructed of PMMA teeth and a visiolign pink composite estimating the gingival tissue.
  Other Names: Titanium prosthesis
Device: Titanium prosthesis — For the TP, the framework will be milled from Ti blocks according to the virtual design of the final prosthesis framework. PMMA teeth then will be cemented, and the final prosthesis will be screwed.

SUMMARY:
This crossover clinical study will examine the impact of the framework material of implant-supported prostheses on patient satisfaction and Oral Health-Related Quality of Life (OHRQoL) with mandibular All-on-4 implant distribution. The trial will investigate subject satisfaction, OHRQoL as the primary outcome, and chewing efficiency and maximum bite force as secondary outcomes for different framework materials used in implant-supported screw-retained restorations. The first null hypothesis states no significant difference in patient satisfaction and OHRQoL between the tested prostheses. Additionally, the second null hypothesis states no significant difference in chewing efficiency and maximum bite force between the tested prostheses.

DETAILED DESCRIPTION:
Prosthetic steps

1. For each patient, an abutment-level impression will be made, and the resultant cast will be 3D scanned for CAD/CAM construction of a PEEK superstructure with abutments.
2. A verification jig will be constructed to ensure the accuracy of the cast.
3. The final prosthesis will be virtually planned by using the Exo-Cad software.
4. The final prosthesis will be milled in Duralay polymerized resin disk, and the prosthesis resin pattern will be tried intra-orally for passive fit using a screw test.
5. For the PP, The PEEK framework will be constructed, the fit of the PEEK framework will be verified intraorally, and the final screw-retained prosthesis will be constructed of PMMA teeth and a visiolign pink composite estimating the gingival tissue.
6. For the TP, the framework will be milled from Ti blocks according to the virtual design of the final prosthesis framework. PMMA teeth then will be cemented, and the final prosthesis will be screwed.

Evaluation

1. Patient satisfaction (VAS) Patient satisfaction will be evaluated using a questionnaire based on a visual analog scale (VAS).(21) Patients will be asked to mark their answer (amount of satisfaction) on a 100-mm line (with zero referring to not satisfied at all and 100 referring to completely satisfied). The mean of the answers (length of the lines from zero to the marks in mm) for each question was subjected to statistical analysis.
2. Oral health-related quality of life (OHIP-14) The oral health impact profile (OHIP-14) questionnaire was used to measure OHRQoL. The full OHIP questionnaire consisted of 49 items covering seven main domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, and social disability. The OHIP-14 questionnaires were translated into Arabic by linguistic professionals who worked in collaboration with the authors to prepare the final version.
3. Evaluation of masticatory efficiency: Chewing efficiency will be evaluated using the color mixing ability test.
4. Evaluation of maximum bite force (BF): A digital BF transducer will be used to evaluate maximum BF in Newton (N).

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria include

* healthy male patients free from systemic diseases that may affect bone health, such as uncontrolled diabetes mellitus and osteoporosis.
* implants placed with the All-on-4 concept in the mandible.

Exclusion Criteria:

* The exclusion criteria: the patients with a history of parafunctional habits (bruxism and clenching), smoking, and alcoholism

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 3 month
  Patient satisfaction will be evaluated using a questionnaire based on a visual analog scale
chewing efficiency | 3 month
  Chewing efficiency will be evaluated using the color mixing ability test

SECONDARY OUTCOMES:
Oral health-related quality of life (OHRQoL) | 3 month
  The oral health impact profile (OHIP-14) questionnaire was used to measure OHRQoL.
maximum bite force (BF) | 3 month
  A digital BF transducer will be used to evaluate maximum BF in Newton (N)

CONTACTS AND LOCATIONS:
Overall Officials: Khloud Ezzat, PhD, Principal Investigator — Lecturer
Locations (1):
- Khloud Ezzat, Al Mansurah, Egypt